CLINICAL TRIAL: NCT05756647
Title: Mandibular Advancement vs Home Treatment for Primary Snoring: A Randomized Trial (SNORE-LESS)
Brief Title: Mandibular Advancement vs Home Treatment for Primary Snoring
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Vice chair for Research Department of Otolaryngology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202208175
Record Dates: First submitted 2023-02-01; First posted 2023-03-06 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Snoring
Keywords: Mandibular Advancement Devices (MAD); external nasal dilator; mouth tapping; lateral positional therapy; Breath-rite strip; Mometasone Nasal Rinse
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial with an active control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: * Due to the nature of the randomization process, blinding during the data collection phase will not be possible.
  * Participants cannot be blinded either as the treatment modalities differ in a way which makes adequate blinding not possible.
  * Prior to data analysis, Dr. Kallogjeri will blind groups as "A" and "B" so that the team will not know which intervention corresponds to A and B throughout both the data analysis and manuscript writing process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional Arm (Experimental): The Mandibular Advancement Device for this study will be the ProSomnus Sleep Device. It is a sleep device intended to reduce nighttime snoring and mild to moderate Obstructive Sleep Apnea in adults by holding the lower jaw forward during sleep
  Interventions: Device: Interventional Arm
- Conservative treatment Arm (Active Comparator): The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Interventions: Combination Product: Conservative treatment Arm

INTERVENTIONS:
Device: Interventional Arm — The MAD arm will consist of participants given a fitted mandibular advancement device that they will wear for the length of the study.
  Other Names: MAD (anti-snoring mouthpiece)
  Arms: Interventional Arm
Combination Product: Conservative treatment Arm — Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
  Arms: Conservative treatment Arm

SUMMARY:
This is a randomized controlled trial for non-apneic snorers. The primary goal of the study is to evaluate the efficacy of a mandibular advancement device (MAD) vs conservative treatment for adults with non-apneic snoring as measured by the partners report of response to treatment (CGI-I). The secondary goal is to evaluate the effectiveness of treatment of snoring on the Epworth Sleepiness Scale (ESS), a modified Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) questionnaire, the Pittsburgh Sleep Quality Index (PSQI), and the Clinical Global Impression of Severity Scale (CGI-S)

DETAILED DESCRIPTION:
Snoring is a problem which affects roughly half of adults, but rigorous studies on how to treat isolated snoring have not been completed. Mandibular advancement devices (MAD) show consistent improvements in sleep quality for patients with sleep apnea; however, their effect on patients with primary snoring remains less well known.

The primary hypothesis proposes that adults with non-apneic snoring treated with a MAD will experience a greater reduction of snoring as measured by the Clinical Global Impression - Improvement (GCI-I) Scale response of the sleeping partner.

The plan is to enroll 30 participants and 30 sleeping partner participants for each arm of the trial: 120 participants, or 60 pairs, in total. Participants will use the intervention nightly for a period of 4 weeks after which an end of study visit will occur. All post intervention outcomes will be recorded at the end of the study visit. Knowledge gained from this study will help guide treatment practice and evidence-based approaches regarding non-apneic snoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Report of snoring
* Prior polysomnogram (PSG) within the past 60 months showing AHI (Apnea Hypopnea Index) < 5 and no more than 10% gain in body weight since the prior polysomnogram OR reasonable clinical suspicion that the participant does not have sleep apnea [Reasonable Clinical Suspicion is defined as: BMI <35, Neck circumference <16.5 inches, lack of uncontrolled hypertension, no witnessed episodes of apnea, or multiple sleep studies in the past all showing lack of sleep apnea but with >5 years since the most recent one.]
* Possess a sleeping partner who sleeps in the same room as the participant for >= 4 nights a week and who can report outcomes
* Access to the internet
* Ability to follow up within 1 month after adequate fitting of MAD or 4 weeks of Mometasone

Inclusion criteria for the sleeping partner:

* Age ≥ 18
* Possess a sleeping partner who sleeps in the same room as the participant for >= 4 nights a week and who can report outcomes
* Access to the internet

Exclusion Criteria:

Individuals will not be allowed to participate in this study if they meet one or more of the exclusion criteria:

* Significant hypoxemia as defined as SaO2 (oxygen saturation) below 89% for ≥ 12% of the total nocturnal monitoring time
* Inability to wear a MAD defined as missing more than 50% of their dentition or their dentition is not in good condition.
* Prior intolerance of MAD
* Current treatment for OSA
* Concurrent use of sedatives or > 2 alcoholic drinks per night
* Chronic nasal obstruction due to structural anatomic defects, nasal polyps, or history of unresponsiveness to nasal rinses.

Sleeping partners do not have any exclusion criteria defined for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffstein V. Snoring. Chest. 1996 Jan;109(1):201-22. doi: 10.1378/chest.109.1.201. No abstract available. PMID 8549187
- [Background] Horner RL. Pathophysiology of obstructive sleep apnea. J Cardiopulm Rehabil Prev. 2008 Sep-Oct;28(5):289-98. doi: 10.1097/01.HCR.0000336138.71569.a2. PMID 18784537
- [Background] Parati G, Lombardi C, Hedner J, Bonsignore MR, Grote L, Tkacova R, Levy P, Riha R, Bassetti C, Narkiewicz K, Mancia G, McNicholas WT; European Respiratory Society; EU COST ACTION B26 members. Position paper on the management of patients with obstructive sleep apnea and hypertension: joint recommendations by the European Society of Hypertension, by the European Respiratory Society and by the members of European COST (COoperation in Scientific and Technological research) ACTION B26 on obstructive sleep apnea. J Hypertens. 2012 Apr;30(4):633-46. doi: 10.1097/HJH.0b013e328350e53b. PMID 22406463
- [Background] Marshall NS, Wong KK, Cullen SR, Knuiman MW, Grunstein RR. Snoring is not associated with all-cause mortality, incident cardiovascular disease, or stroke in the Busselton Health Study. Sleep. 2012 Sep 1;35(9):1235-40. doi: 10.5665/sleep.2076. PMID 22942501
- [Background] Jennum P, Hein HO, Suadicani P, Gyntelberg F. Risk of ischemic heart disease in self-reported snorers. A prospective study of 2,937 men aged 54 to 74 years: the Copenhagen Male Study. Chest. 1995 Jul;108(1):138-42. doi: 10.1378/chest.108.1.138. PMID 7606948
- [Background] Hoffstein V. Blood pressure, snoring, obesity, and nocturnal hypoxaemia. Lancet. 1994 Sep 3;344(8923):643-5. doi: 10.1016/s0140-6736(94)92084-2. PMID 7915347
- [Background] Yeboah J, Redline S, Johnson C, Tracy R, Ouyang P, Blumenthal RS, Burke GL, Herrington DM. Association between sleep apnea, snoring, incident cardiovascular events and all-cause mortality in an adult population: MESA. Atherosclerosis. 2011 Dec;219(2):963-8. doi: 10.1016/j.atherosclerosis.2011.08.021. Epub 2011 Aug 22. PMID 22078131
- [Background] Deeb R, Smeds MR, Bath J, Peterson E, Roberts M, Beckman N, Lin JC, Yaremchuk K. Snoring and carotid artery disease: A new risk factor emerges. Laryngoscope. 2019 Jan;129(1):265-268. doi: 10.1002/lary.27314. Epub 2018 Sep 8. PMID 30194704
- [Background] Lee SA, Amis TC, Byth K, Larcos G, Kairaitis K, Robinson TD, Wheatley JR. Heavy snoring as a cause of carotid artery atherosclerosis. Sleep. 2008 Sep;31(9):1207-13. PMID 18788645
- [Background] Jennum P, Hein HO, Suadicani P, Gyntelberg F. Cognitive function and snoring. Sleep. 1993 Dec;16(8 Suppl):S62-4. doi: 10.1093/sleep/16.suppl_8.s62. PMID 8178029
- [Background] Parish JM, Lyng PJ. Quality of life in bed partners of patients with obstructive sleep apnea or hypopnea after treatment with continuous positive airway pressure. Chest. 2003 Sep;124(3):942-7. doi: 10.1378/chest.124.3.942. PMID 12970021
- [Background] Beninati W, Harris CD, Herold DL, Shepard JW Jr. The effect of snoring and obstructive sleep apnea on the sleep quality of bed partners. Mayo Clin Proc. 1999 Oct;74(10):955-8. doi: 10.4065/74.10.955. PMID 10918859
- [Background] Troxel WM, Buysse DJ, Hall M, Matthews KA. Marital happiness and sleep disturbances in a multi-ethnic sample of middle-aged women. Behav Sleep Med. 2009;7(1):2-19. doi: 10.1080/15402000802577736. PMID 19116797
- [Background] Blumen MB, Quera Salva MA, Vaugier I, Leroux K, d'Ortho MP, Barbot F, Chabolle F, Lofaso F. Is snoring intensity responsible for the sleep partner's poor quality of sleep? Sleep Breath. 2012 Sep;16(3):903-7. doi: 10.1007/s11325-011-0554-5. Epub 2011 Jul 10. PMID 21744233
- [Background] Patel M, Tran D, Chakrabarti A, Vasquez A, Gilbert P, Davidson T. Prevalence of snoring in college students. J Am Coll Health. 2008 Jul-Aug;57(1):45-52. doi: 10.3200/JACH.57.1.45-52. PMID 18682345
- [Background] Rich J, Raviv A, Raviv N, Brietzke SE. An epidemiologic study of snoring and all-cause mortality. Otolaryngol Head Neck Surg. 2011 Aug;145(2):341-6. doi: 10.1177/0194599811402475. PMID 21493281
- [Background] Braver HM, Block AJ. Effect of nasal spray, positional therapy, and the combination thereof in the asymptomatic snorer. Sleep. 1994 Sep;17(6):516-21. doi: 10.1093/sleep/17.6.516. PMID 7528939
- [Background] Nakano H, Ikeda T, Hayashi M, Ohshima E, Onizuka A. Effects of body position on snoring in apneic and nonapneic snorers. Sleep. 2003 Mar 15;26(2):169-72. doi: 10.1093/sleep/26.2.169. PMID 12683476
- [Background] Cartwright R, Ristanovic R, Diaz F, Caldarelli D, Alder G. A comparative study of treatments for positional sleep apnea. Sleep. 1991 Dec;14(6):546-52. doi: 10.1093/sleep/14.6.546. PMID 1798889
- [Background] De Meyer MMD, Vanderveken OM, De Weerdt S, Marks LAM, Carcamo BA, Chavez AM, Matamoros FA, Jacquet W. Use of mandibular advancement devices for the treatment of primary snoring with or without obstructive sleep apnea (OSA): A systematic review. Sleep Med Rev. 2021 Apr;56:101407. doi: 10.1016/j.smrv.2020.101407. Epub 2020 Nov 29. PMID 33326914
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Smith SS, Oei TP, Douglas JA, Brown I, Jorgensen G, Andrews J. Confirmatory factor analysis of the Epworth Sleepiness Scale (ESS) in patients with obstructive sleep apnoea. Sleep Med. 2008 Oct;9(7):739-44. doi: 10.1016/j.sleep.2007.08.004. Epub 2007 Oct 24. PMID 17921053
- [Background] Piccirillo JF. Outcomes research and obstructive sleep apnea. Laryngoscope. 2000 Mar;110(3 Pt 3):16-20. doi: 10.1097/00005537-200003002-00005. PMID 10718409
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Brown HJ, Batra PS, Eggerstedt M, Ganti A, Papagiannopoulos P, Tajudeen BA. The possibility of short-term hypothalamic-pituitary-adrenal axis suppression with high-volume, high-dose nasal mometasone irrigation in postsurgical patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2022 Mar;12(3):249-256. doi: 10.1002/alr.22894. Epub 2021 Sep 26. PMID 34569177
- [Background] Jiramongkolchai P, Peterson A, Kallogjeri D, Lee JJ, Kukuljan S, Liebendorfer A, Schneider JS, Klatt-Cromwell CN, Drescher AJ, Piccirillo JF. Randomized clinical trial to evaluate mometasone lavage vs spray for patients with chronic rhinosinusitis without nasal polyps who have not undergone sinus surgery. Int Forum Allergy Rhinol. 2020 Aug;10(8):936-943. doi: 10.1002/alr.22586. Epub 2020 May 29. PMID 32470217
- [Derived] Ioerger P, Afshari A, Hentati F, Strober W, Kallogjeri D, Ju YE, Piccirillo JF. Mandibular Advancement vs Combined Airway and Positional Therapy for Snoring: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Jul 1;150(7):572-579. doi: 10.1001/jamaoto.2024.1035. PMID 38780959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We only enrolled 100 study participants.
Groups:
- Interventional Arm: Snorers; Interventional Arm: Partners: The Mandibular Advancement Device for this study will be the ProSomnus Sleep Device. It is a sleep device intended to reduce nighttime snoring and mild to moderate Obstructive Sleep Apnea in adults by holding the lower jaw forward during sleep
  Interventional Arm: The MAD arm will consist of participants given a fitted mandibular advancement device that they will wear for the length of the study.
- Conservative Treatment Arm: Snorers; Conservative Arm: Partners: The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Conservative treatment Arm: Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
Period: Overall Study
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm: Partners | Conservative Arm: Partners
Started (A total of 100 study participants were enrolled in the study.) | 25 | 25 | 25 | 25
Completed | 23 | 19 | 23 | 19
Not Completed | 2 | 6 | 2 | 6

BASELINE CHARACTERISTICS:
Population: We enrolled snoring individuals and their sleeping partners.
Groups:
- Conservative Treatment Arm: Partners: The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Conservative treatment Arm: Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
- Total: Total of all reporting groups
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm: Partners | Conservative Treatment Arm: Partners | Total
Number analyzed (Participants) | 23 | 19 | 23 | 19 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.8) | 45.5 (14.4) | 47.1 (16.8) | 43.0 (16.2) | 47.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Characteristics for snoring and sleeping partners were reported in dyads.
  Participants
    Female | 15 | 11 | 10 | 9 | 45
    Male | 8 | 8 | 13 | 10 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 22 | 19 | 20 | 18 | 79
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
CGI-S [Count of Participants; unit: Participants] — Population: Response options for the CGI-S were none, mild, moderate, severe, and problem as bad as it can be. Participants who rated the snoring as mild, moderate, severe, or problem as bad as it can be were defined as problematic snoring.
  Participants
    None | 0 | 1 | 2 | 0 | 3
    Mild | 8 | 9 | 3 | 7 | 27
    Moderate | 12 | 7 | 9 | 6 | 34
    Severe | 3 | 2 | 9 | 5 | 19
    As bad as it can be | 0 | 0 | 0 | 1 | 1
ESS [Median (Full Range); unit: score on a scale 0-24] — The ESS is a commonly used measure to evaluate the propensity to of a participant to fall asleep in 8 everyday scenarios "in recent times". The participant rates each situation on a scale of 1-7, with 1 being least likely to fall asleep and 7 being the most likely.
  The total score for the Epworth Sleepiness Scale (ESS) ranges from 0 to 24, with higher scores indicating greater daytime sleepiness, and a score of 10 or greater suggesting excessive daytime sleepiness.
  score on a scale 0-24 | 4 [0 to 16] | 6 [2 to 14] | 4 [0 to 12] | 6 [0 to 14] | 4.5 [0 to 16]
PSQI [Median (Full Range); unit: score on a scale 0-21] — The PSQI is a self-rate questionnaire which assess sleep quality and disturbances over a 1- month time interval. It is composed of 19 items which contribute to 7 different component scores.
  The total score for the Pittsburgh Sleep Quality Index (PSQI) ranges from 0 to 21, with higher scores indicating poorer sleep quality.
  score on a scale 0-21 | 6 [1 to 17] | 7 [3 to 16] | 6 [2 to 14] | 6 [3 to 18] | 7 [1 to 17]
SNORE-25 [Median (Full Range); unit: score on a scale 0-5] — The SNORE-25 is a modification of the Obstructive Sleep Apnea Patient-Oriented Severity Index (OSAPOSI) which includes 25 total items of symptoms with possible scores ranging from 0 to 5, with high scores indicating greater sleep-disordered breathing-related health burden.
  score on a scale 0-5 | 0.48 [0.08 to 1.8] | 1.20 [0.28 to 2.08] | 1 [0.1 to 2.2] | 1.04 [0.2 to 2.16] | 0.72 [0.08 to 2.08]

OUTCOME MEASURES:

1. Primary Outcome: Percent Responders of Clinical Global Impression of Improvement Scale - Partner
Description: This will occur asynchronously through email surveys distributed through the Washington University REDCap server or through a scheduled telephone call depending on the participant's preference. The Partner will grade the improvement of the snoring on the following continuous scale, which will be the Clinical Global Impression of Improvement (CGI-I) scale:
  Very Much Improved Much Improved Minimally Improved No Change Minimally Worse Much Worse Very Much Worse
  The percentage of responders to treatment will then be compared between the two arms of the trial. A responder will be defined as someone who rates the response to snoring as either "Very Much Improved" or "Much Improved"
Time Frame: 4 weeks post intervention beginning
Measure: Number; unit: percent of snorer responders
Arm/Group | Interventional Arm | Conservative Treatment Arm
Number analyzed (Participants) | 21 | 11
percent of snorer responders | 91 | 58

2. Secondary Outcome: Change in Clinical Global Impression of Severity Scale
Description: The CGI-Severity Scale poses the question "On average, how much of a problem does your [partner's] snoring pose?" The 5 response options will include: no problem, mild problem, moderate problem, severe problem, problem as severe as it can be. It will be measured both at baseline and after treatment. Change in CGI-S score will be calculated and reported as a secondary outcome measure as the change in CGI-S score between the two arms. In addition, the CGI-S will be measured by the sleeping partner on a daily basis both before and after treatment.
Time Frame: 4 weeks post intervention beginning
Measure: Number; unit: responders
Groups:
- Interventional Arm: Snorer; Interventional Arm: Partner: The Mandibular Advancement Device for this study will be the ProSomnus Sleep Device. It is a sleep device intended to reduce nighttime snoring and mild to moderate Obstructive Sleep Apnea in adults by holding the lower jaw forward during sleep
  Interventional Arm: The MAD arm will consist of participants given a fitted mandibular advancement device that they will wear for the length of the study.
- Conservative Treatment Arm: Snorer; Conservative Treatment Arm: Partner: The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Conservative treatment Arm: Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
Arm/Group | Interventional Arm: Snorer | Conservative Treatment Arm: Snorer | Interventional Arm: Partner | Conservative Treatment Arm: Partner
Number analyzed (Participants) | 23 | 19 | 23 | 19
responders
  None | 6 | 2 | 9 | 2
  Mild | 8 | 8 | 8 | 9
  Moderate | 7 | 7 | 4 | 6
  Severe | 2 | 2 | 2 | 1
  As bad as it can be | 0 | 0 | 0 | 1

3. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) Score
Description: The ESS is a commonly used measure to evaluate the propensity to of a participant to fall asleep in 8 everyday scenarios "in recent times". The participant rates each situation on a scale of 0-3, with 0 being least likely to fall asleep and 3 being the most likely. Final score can range from 0-24. Epworth Sleepiness Scale (ESS) score will be recorded by both the partner and the snorer at baseline and follow up. Change in ESS score will be calculated and reported as a secondary outcome measure as the change in ESS score or the difference in percentage of participates recording an ESS improvement above the Minimal Clinically Important Difference between the two arms.
Time Frame: Baseline and 4 weeks post intervention beginning
Measure: Median (Full Range); unit: score on a scale
Groups:
- Conservative Treatment Arm:Partners: The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Conservative treatment Arm: Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm: Partners | Conservative Treatment Arm:Partners
Number analyzed (Participants) | 23 | 19 | 23 | 19
score on a scale | 2 [0 to 13] | 4 [0 to 14] | 4 [0 to 12] | 6 [0 to 14]

4. Secondary Outcome: Change in Symptoms of Nocturnal Obstruction and Related Events (SNORE-25)
Description: The SNORE-25 is a modification of the Obstructive Sleep Apnea Patient-Oriented Severity Index (OSAPOSI) which includes 25 total items. Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) score will be recorded by both the partner and the snorer at baseline and follow up.
  The SNORE-25 score is calculated as the mean item score for all 25 items. The possible range for the SNORE-25 score is 0-5, with higher scores indicating greater sleep disordered-related health burden.
  Impact of treatment is assessed with the SNORE-25 Change Score.
  The SNORE-25 Change Score is the difference between SNORE-25 Pre-treatment and SNORE-25 Post-Treatment scores.
  Minimal Clinically Important Difference. A SNORE-25 Change Score of 0.5 should be considered the minimal clinically important difference and change scores greater than this should be considered clinically meaningful.
Time Frame: Baseline and 4 weeks post intervention beginning
Population: Comparison of outcome measures between the study group
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm: Partners | Conservative Treatment Arm: Partners
Number analyzed (Participants) | 23 | 19 | 23 | 19
score on a scale | 0.2 [0.04 to 1.6] | 0.54 [0.12 to 1.84] | 0.2 [0.04 to 2.04] | 0.88 [0.04 to 2.48]

5. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index is a self-rate questionnaire which assess sleep quality and disturbances over a 1-month time interval. It is composed of 19 items which contribute to 7 different component scores:A global sum of these components > 5 signifies poor sleep quality with a sensitivity of 89.6% and a specific of 86.5%2
  Change in Pittsburgh Sleep Quality Index score will be calculated and reported as a secondary outcome measure as the change in Pittsburgh Sleep Quality Index score or the difference in percentage of participates recording a Pittsburgh Sleep Quality Index improvement above the Minimal Clinically Important Difference (4.4) compared between the two arms.
  The questionnaire consists of a combination of Likert type and open-ended questions (later converted to scaled scores).Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Time Frame: Baseline and follow up
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm: Partners | Conservative Treatment Arm: Partners
Number analyzed (Participants) | 23 | 19 | 23 | 19
score on a scale | 2 [1 to 10] | 4 [1 to 10] | 4 [1 to 12] | 6 [1 to 17]

6. Secondary Outcome: Percent Responder of Clinical Global Impression of Improvement Scale - Snorer
Description: The Snorer will grade the improvement of their own snoring on the following scale, which will be the Clinical Global Impression of Improvement (CGI-I) scale:
  Very Much Improved Much Improved Minimally Improved No Change Minimally Worse Much Worse Very Much Worse
  The percentage of responders to treatment will then be compared between the two arms of the trial. A responder will be defined as someone who rates the response to snoring as either "Very Much Improved" or "Much Improved"
Time Frame: 4 weeks post intervention beginning
Measure: Number; unit: percentage of responders
Groups:
- Interventional Arm - Snorer; Interventional Arm - Partner: The Mandibular Advancement Device for this study will be the ProSomnus Sleep Device. It is a sleep device intended to reduce nighttime snoring and mild to moderate Obstructive Sleep Apnea in adults by holding the lower jaw forward during sleep
  Interventional Arm: The MAD arm will consist of participants given a fitted mandibular advancement device that they will wear for the length of the study.
- Conservative Treatment Arm- Snorer; Conservative Treatment Arm - Partner: The conservative treatment will consist of four different interventions: Mometasone nasal rinse, External nasal dilatory therapy, Mouth taping and Lateral positional therapy.
  Conservative treatment Arm: Participant will undergo a nightly medicated nasal rinse that will occur for a 4 week period, prior to beginning of the other three conservative therapy interventions. The 4-part combination therapy will take place for 4 weeks total.
Arm/Group | Interventional Arm - Snorer | Conservative Treatment Arm- Snorer | Interventional Arm - Partner | Conservative Treatment Arm - Partner
Number analyzed (Participants) | 21 | 8 | 21 | 11
percentage of responders | 91 | 44 | 91 | 58

ADVERSE EVENTS:
Time Frame: Serious adverse events (within 1week) Any other problems ( within 2 weeks) Intervention treatment time frame was 4 weeks.
Description: No serious adverse events were reported. There were no participants at risk for all cause mortality.
Groups:
- Interventional Arm:Partners: The Mandibular Advancement Device for this study will be the ProSomnus Sleep Device. It is a sleep device intended to reduce nighttime snoring and mild to moderate Obstructive Sleep Apnea in adults by holding the lower jaw forward during sleep
  Interventional Arm: The MAD arm will consist of participants given a fitted mandibular advancement device that they will wear for the length of the study.
Arm/Group | Interventional Arm: Snorers | Conservative Treatment Arm: Snorers | Interventional Arm:Partners | Conservative Treatment Arm:Partners
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19 | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19 | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 10/23 | 5/19 | 0/23 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm: Snorers (N=23) | Conservative Treatment Arm: Snorers (N=19) | Interventional Arm:Partners (N=23) | Conservative Treatment Arm:Partners (N=19)
Jaw pain (General disorders) | 10 (10) | 0 (0) | 0 (0) | 0 (0) — reported self-resolving jaw pain/discomfort for a few days after beginning the device.
sinus headache (General disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) — Brief "sinus headache" upon starting the nasal saline rinse.
Unable to tolerate side effects of the treatment (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — pre treatment
Unable tolerate the side effects of the treatment (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — during treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT05756647/Prot_SAP_000.pdf